CLINICAL TRIAL: NCT04345601
Title: Single Donor Banked Bone Marrow Mesenchymal Stromal Cells for the Treatment of COVID-19 Induced ARDS: A Non-Blinded Randomized, Controlled Study
Brief Title: Mesenchymal Stromal Cells for the Treatment of SARS-CoV-2 Induced Acute Respiratory Failure (COVID-19 Disease)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, LaQuisa Hill, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-47561 MSC for COVID-19
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Results first posted 2024-04-01 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Sars-CoV2; Acute Respiratory Distress Syndrome; COVID-19
Keywords: Mesenchymal Stromal Cells; Respiratory failure
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19; Respiratory Insufficiency | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Safety Run In (Experimental): The study will first enroll and treat six patients with MSCs for safety run in. If no more than 2 treatment-related severe adverse events (tSAEs) are observed, the study will enroll and randomize additional patients in a ratio of 1:1 to receive either MSCs or routine/supportive care.
  Interventions: Biological: Mesenchymal Stromal Cells
- Mesenchymal stromal cells (Experimental): Patients randomized to the MSC arm will be administered an intravenous infusion of MSCs at a dose of 1 x 10^8. A second infusion will be allowed if the patient does not have improvement in respiratory parameters per discretion of the investigator, or ARDS clinically worsens, within 3-5 days following the initial infusion.
  Interventions: Biological: Mesenchymal Stromal Cells
- Control Group (Other): Patients randomized to the control arm will receive supportive care or treatment designated by their treating physicians.
  Interventions: Other: Supportive Care

INTERVENTIONS:
Biological: Mesenchymal Stromal Cells — Patients will be given the cell product by intravenous injection (into the vein through an IV line). Dose:1 x 10^8 MSCs.
  Other Names: MSCs
  Arms: Mesenchymal stromal cells; Safety Run In
Other: Supportive Care — Patients will receive supportive care per their treating physician
  Arms: Control Group

SUMMARY:
***At this time, we are only enrolling at Houston Methodist Hospital (HMH)/Baylor College of Medicine (BCM) and are not shipping cells outside of BCM/HMH.***

This is a study for patients who have respiratory infection caused by SARS-CoV-2 that have not gotten better. Because there is no standard treatment for this infection, patients are being asked to volunteer for a gene transfer research study using mesenchymal stem cells (MSCs).

Stem cells are cells that do not yet have a specific function in the body. Mesenchymal stem cells (MSCs) are a type of stem cell that can be grown from bone marrow (the spongy tissue inside of bones). Stem cells can develop into other types of more mature (specific) cells, such as blood and muscle cells.

The purpose of this study is to see if MSCs versus controls can help to treat respiratory infections caused by SARS-CoV-2.

DETAILED DESCRIPTION:
Earlier, a healthy donor provided blood cells to generate MSCs. These cells were grown and frozen for later use.

Before being treated, the patient will receive a series of standard medical tests: These tests are done to assess the patient's eligibility to receive the cells.

* Physical exam and history
* SARS-CoV-2 test
* Blood tests
* Chest X-ray or chest CT Scan
* A urine pregnancy test, when applicable

The patient will be randomly assigned to a study group. We'll use a computer to put the patient into study group A (study drug) or group B (control) by chance (randomized). Patients randomized to the control group, will receive the standard treatment for their respiratory infection.

On the day that the patient is scheduled to receive the cells they will be pre-medicated with Benadryl and Tylenol. The patient will then receive an intravenous (into the vein) infusion of 1 x 10^8 cells/kg of MSCs. The patient will be monitored closely for two hours after the infusion. The patient will receive a second infusion at the same dose within 3-5 days of the initial infusion (at the discretion of the investigator) if there is no improvement in respiratory parameters or if there is a worsening of Acute respiratory distress syndrome (ARDS).

The patient will receive standard medical tests when getting the infusion(s) and afterwards. As part of the research study, the patient will be evaluated daily for 7 days and then weekly at weeks 2, 3, and 4. The evaluations that will be done at these visits include:

* Physical exam and history
* SARS-CoV-2 test
* Blood tests
* Chest X-ray or chest CT Scan

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Confirmed SARS-CoV2 infection real-time reverse transcription polymerase chain reaction (RT-PCR) assay
3. Moderate OR severe ARDS, based on the degree of impairment of oxygenation as defined by the ratio of arterial oxygen tension to fraction of inspired oxygen (PaO2/FiO2):

   1. Moderate ARDS: PaO2/FiO2 100-200 mmHg OR
   2. Severe ARDS: PaO2/FiO2 ≤100 mmHg
4. If on invasive or noninvasive (BiPAP) mechanical ventilator, PEEP ≥5 cm H2O
5. Bilateral opacities present on chest radiograph or computed tomographic (CT) scan, that are not fully explained by pleural effusions, lung collapse, or lung nodules.

Exclusion Criteria:

1. Currently receiving extracorporeal membrane oxygenation (ECMO)
2. Severe chronic respiratory disease requiring use of home oxygen
3. Pregnant or lactating
4. Known hypersensitivity to dimethyl sulfoxide (DMSO)
5. Unstable hemodynamics as deemed by the treating physician/investigator including but not limited to unstable, ventricular tachycardia or new cardiac arrythmia requiring cardioversion.
6. Uncontrolled bacterial or fungal co-infection
7. Any end-stage organ disease or condition, which in the opinion of the Investigator, makes the patient an unsuitable candidate for treatment
8. Inability to obtain informed consent (from patient or legally appropriate proxy)
9. Presence of any contraindication to receiving prophylactic low dose unfractionated or low molecular weight heparin.
10. Respiratory failure not fully explained by cardiac failure or fluid overload.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: LaQuisa Hill, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Safety Run In: The study will first enroll and treat six patients with mesenchymal stromal cells(MSCs) for safety run in. If no more than 2 treatment-related severe adverse events (tSAEs) are observed, the study will enroll and randomize additional patients in a ratio of 1:1 to receive either MSCs or routine/supportive care.
  Mesenchymal Stromal Cells(MSCs): Patients will be given the cell product by intravenous injection (into the vein through an IV line). Dose:1 x 10^8 MSCs.
- Mesenchymal Stromal Cells (MSCs): Patients randomized to the MSC arm will be administered an intravenous infusion of MSCs at a dose of 1 x 10^8. A second infusion will be allowed if the patient does not have improvement in respiratory parameters per discretion of the investigator, or acute respiratory distress syndrome (ARDS) clinically worsens, within 3-5 days following the initial infusion.
  Mesenchymal Stromal Cells (MSCs): Patients will be given the cell product by intravenous injection (into the vein through an IV line). Dose:1 x 10^8 MSCs.
Period: Overall Study
Arm/Group | Safety Run In | Mesenchymal Stromal Cells (MSCs) | Control Group
Started | 6 | 10 | 12
Completed | 6 | 7 | 8
Not Completed | 0 | 3 | 4
Not completed — Death | 0 | 3 | 2
Not completed — Lost to Follow-up | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Safety Run In: The study will first enroll and treat six patients with mesenchymal stromal cells (MSCs) for safety run in. If no more than 2 treatment-related severe adverse events (tSAEs) are observed, the study will enroll and randomize additional patients in a ratio of 1:1 to receive either MSCs or routine/supportive care.
  Mesenchymal Stromal Cells(MSCs): Patients will be given the cell product by intravenous injection (into the vein through an IV line). Dose:1 x 10^8 MSCs.
- Mesenchymal Stromal Cells (MSCs): Patients randomized to the MSC arm will be administered an intravenous infusion of MSCs at a dose of 1 x 10^8. A second infusion will be allowed if the patient does not have improvement in respiratory parameters per discretion of the investigator, or ARDS clinically worsens, within 3-5 days following the initial infusion.
  Mesenchymal Stromal Cells(MSCs): Patients will be given the cell product by intravenous injection (into the vein through an IV line). Dose:1 x 10^8 MSCs.
- Total: Total of all reporting groups
Arm/Group | Safety Run In | Mesenchymal Stromal Cells (MSCs) | Control Group | Total
Number analyzed (Participants) | 6 | 10 | 12 | 28
Age, Continuous [Median (Full Range); unit: years] | 58.5 [40 to 64] | 56.5 [27 to 74] | 52.0 [38 to 72] | 55 [27 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 5 | 12
  Male | 2 | 7 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 4 | 11
  Not Hispanic or Latino | 4 | 4 | 7 | 15
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 3
  White | 5 | 9 | 9 | 23
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Treatment-related Serious Adverse Events (tSAEs)
Description: Treatment-related serious adverse events (tSAE) are those directly related to the investigational infusion product. Adverse event grading will be per NCI Common Terminology Criteria for Adverse Events(CTCAE), vs 5. Rate of tSAEs in patients treated with MSCs will be reported as proportion and its 95% confidence interval.
Time Frame: 28 days post cell infusion
Population: All participants who received MSCs are included in the analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participant
Arm/Group | Safety Run In | Mesenchymal Stromal Cells | Control Group
Number analyzed (Participants) | 6 | 10 | 0
proportion of participant | 0 [0 to 0.4593] | 0 [0 to 0.3085] |

2. Primary Outcome: Number of Participants With Improvement by at Least Two Categories on a Six Category Ordinal Scale at Day 14
Description: Change by at least two categories on a six-category ordinal scale as improvement at day 14 post-randomization per protocol defined criteria. The six-category ordinal scale ranges from 6 to 1 with a higher score indicating a worse clinical outcome as follows: 6 ꞊ death; 5 ꞊ hospitalization, requiring extracorporeal membrane oxygenation (ECMO) and/or invasive mechanical ventilation (IMV); 4 ꞊ hospitalization, requiring non-invasive mechanical ventilation (NIV) and/or High-flow nasal cannula (HFNC) therapy; 3 = hospitalization, requiring supplemental oxygen (but not NIV/HFNC); 2 = hospitalization, not requiring supplemental oxygen; 1 = hospital discharge.
Time Frame: 14 days post cell infusion
Population: All study participants are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Run In | Mesenchymal Stromal Cells | Control Group
Number analyzed (Participants) | 6 | 10 | 12
Participants
  Improved by at least two categories | 2 | 2 | 5
  Not improved by at least two categories | 4 | 8 | 7

3. Secondary Outcome: Clinical Status Determined by 6-point Ordinal Scale at Day 28
Description: Clinical status at day 28 as determined by 6-point ordinal scale as follows: 6 ꞊ death; 5 ꞊ hospitalization, requiring extracorporeal membrane oxygenation (ECMO) and/or invasive mechanical ventilation (IMV); 4 ꞊ hospitalization, requiring non-invasive mechanical ventilation (NIV) and/or High-flow nasal cannula (HFNC) therapy; 3 = hospitalization, requiring supplemental oxygen (but not NIV/HFNC); 2 = hospitalization, not requiring supplemental oxygen; 1 = hospital discharge. The six-category ordinal scale ranges from 6 to 1 with a higher score indicating a worse clinical outcome.
Time Frame: 28 days post cell infusion
Population: All study participants are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Run In | Mesenchymal Stromal Cells | Control Group
Number analyzed (Participants) | 6 | 10 | 12
Participants
  1= hospital discharge | 3 | 4 | 7
  2=hospitalization, not requiring supplemental oxygen | 0 | 0 | 0
  3=hospitalization, requiring supplemental oxygen | 1 | 1 | 2
  4=hospitalization, requiring NIV and/or HFNC therapy | 2 | 0 | 0
  5=hospitalization, requiring ECOM and/or IMV | 0 | 2 | 1
  6=dead | 0 | 3 | 2

4. Secondary Outcome: Severity of Acute Respiratory Distress Syndrome (ARDS) at Day 14
Description: ARDS is divided into 3 groups based on the degree of hypoxemia: mild (partial pressure of oxygen in the arterial blood(PaO2)/fraction of inspired oxygen(FIO2) 201-300 mm Hg), moderate (PaO2/FIO2: 101-200 mm Hg), and severe (PaO2/FIO2 ≤ 100 mm Hg) and ventilator settings with a positive end-expiratory pressure (PEEP) or continuous positive airway pressure (CPAP) ≥5 cm water (H2O).
Time Frame: 14 days post cell infusion
Population: All study participants are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Run In | Mesenchymal Stromal Cells | Control Group
Number analyzed (Participants) | 6 | 10 | 12
Participants
  No ARDS | 1 | 3 | 4
  Mild | 2 | 1 | 2
  Moderate | 2 | 5 | 3
  Severe | 1 | 1 | 3

5. Secondary Outcome: Number of Oxygenation Free Days at Day 28
Description: Number of oxygen support-free days through Day 28
Time Frame: 28 days post cell infusion
Population: All study participants are included in the analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Safety Run In | Mesenchymal Stromal Cells | Control Group
Number analyzed (Participants) | 6 | 10 | 12
days | 6 [0 to 25] | 0 [0 to 21] | 7 [0 to 24]

6. Secondary Outcome: Number of Participants With Progression to Mechanical Ventilation or ECMO
Description: Participants not receiving mechanical ventilation at baseline who progress to requiring mechanical ventilation.
Time Frame: 28 days post cell infusion
Population: Participants who were not receiving mechanical ventilation at baseline are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Run In | Mesenchymal Stromal Cells | Control Group
Number analyzed (Participants) | 5 | 8 | 8
Participants
  Progression to mechanical ventilation or ECMO | 1 | 6 | 3
  No progression to mechanical ventilation or ECMO | 4 | 2 | 5

7. Secondary Outcome: Duration of Mechanical Ventilation and/or ECMO
Description: Number of days requiring invasive mechanical ventilation and/or ECMO (ventilation/ECMO free days at day 28)
Time Frame: 28 days post cell infusion
Population: All participants are included in the analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Safety Run In | Mesenchymal Stromal Cells | Control Group
Number analyzed (Participants) | 6 | 10 | 12
days | 0 [0 to 7] | 11 [0 to 28] | 1 [0 to 20]

8. Secondary Outcome: Duration of ICU Stay
Description: The number of days a participant spent in ICU. Duration of ICU stay is calculated from the date of admission or data of on study if the patient was admitted to ICU before enrollment to the time of ICU discharge, death, or last follow-up, whichever occurred first.
Time Frame: from the date of admission or data of on study if the patient was admitted to ICU before enrollment to the time of ICU discharge, death, or last follow-up, whichever occurred first. Up to 35 days.
Population: Participants admitted to ICU are included in the analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Safety Run In | Mesenchymal Stromal Cells | Control Group
Number analyzed (Participants) | 6 | 9 | 11
days | 16 [4 to 29] | 19 [7 to 35] | 13 [1 to 28]

9. Secondary Outcome: Duration of Hospital Stay
Description: Duration of hospital stay is calculated from the date of on study to the time of hospital discharge, death, or last follow-up, whichever occurred first. It does not reflect the entire hospitalization time.
Time Frame: from the date of on study to the time of hospital discharge, death, or last follow-up, whichever occurred first. Up to 35 days.
Population: All study participants are included in the analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Safety Run In | Mesenchymal Stromal Cells | Control Group
Number analyzed (Participants) | 6 | 10 | 12
days | 24 [4 to 34] | 24 [8 to 35] | 17 [1 to 28]

10. Secondary Outcome: Overall Survival
Description: Probability of overall survival is calculated using Kaplan-Meier survival curves per protocol. Overall survival time is defined as days from the date of randomization or date of infusion if received MSCs to the date of death or the date of the last follow-up for censoring.
Time Frame: 28 days post cell infusion
Population: All study participants are included in the analysis.
Measure: Number (95% Confidence Interval); unit: probability of overall survival
Arm/Group | Safety Run In | Mesenchymal Stromal Cells | Control Group
Number analyzed (Participants) | 6 | 10 | 12
probability of overall survival | 1 [1 to 1] | 0.70 [0.329 to 0.892] | 0.825 [0.461 to 0.953]

11. Secondary Outcome: All-cause Mortality
Description: Number and percentage of deaths (all-cause) until Day 28
Time Frame: 28 days post cell infusion
Population: All study participants are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Run In | Mesenchymal Stromal Cells | Control Group
Number analyzed (Participants) | 6 | 10 | 12
Participants | 0 | 3 | 2

ADVERSE EVENTS:
Time Frame: 28 days after the last dosing of study drug/biologic or until the time of discharge, whichever comes first.
Description: Adverse events are collected as per protocol for participants who received MSCs. All new adverse experiences/toxicities and worsening of baseline toxicities by at least one grade following infusion are collected for 4 weeks after the last dosing of the study drug except for toxicities related to the MSC infusion, which are followed until resolved. Serious Adverse events are collected until 28 days after the last dosing of the study drug or until the time of discharge, whichever comes first.
Arm/Group | Safety Run In | Mesenchymal Stromal Cells (MSCs) | Control Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 3/10 | 2/12
Serious Adverse Events (participants affected / at risk) | 0/6 | 3/10 | 0/12
Other Adverse Events (participants affected / at risk) | 6/6 | 10/10 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Run In (N=6) | Mesenchymal Stromal Cells (MSCs) (N=10) | Control Group (N=12)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Run In (N=6) | Mesenchymal Stromal Cells (MSCs) (N=10) | Control Group (N=12)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4) | 6 (6) | 7 (7)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 10 (10) | 10 (10)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 6 (6) | 4 (5)
Asystole (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Blood bicarbonate decreased (Investigations) | 2 (2) | 7 (7) | 4 (4)
Blood bilirubin increased (Investigations) | 3 (3) | 5 (5) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
CPK increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 4 (4) | 4 (4)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 6 (6) | 5 (5)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fungemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Glucosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 2 (2)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 2 (2)
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (3) | 5 (5) | 4 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 6 (6)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 5 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 7 (7) | 3 (3)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 3 (3)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
INR increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 4 (7)
Lymphocyte count decreased (Investigations) | 2 (2) | 2 (2) | 8 (8)
Metabolism and nutrition disorders - Other, specify:Mild protein-calorie malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 4 (4) | 5 (5) | 7 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify:Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify:rash - unspecified (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Vascular disorders - Other, specify:DVT (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
White blood cell decreased (Investigations) | 0 (0) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/01/NCT04345601/Prot_SAP_001.pdf
  • Informed Consent Form (2022-10-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT04345601/ICF_000.pdf